CLINICAL TRIAL: NCT02719886
Title: Timing of Serial UltrasouNds in High-Risk Pregnancies: A Randomized Controlled Trial
Brief Title: Timing of Serial Ultrasounds
Acronym: SUN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Robyn Roberts, Fellow, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: HSC-MS-15-0968
Record Dates: First submitted 2016-02-11; First posted 2016-03-25 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-12

CONDITIONS: Interval Growth Ultrasound
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fetal growth ultrasound every 2 weeks (Experimental): Ultrasound to measure fetal growth every 2 weeks (i.e. 28, 30, 32, 34, 36, 38 weeks gestation).
  Interventions: Device: Ultrasound
- Fetal growth ultrasound every 4 weeks (Active Comparator): Ultrasound to measure fetal growth every 4 weeks (i.e. 28, 32 and 36 weeks gestation). Usual Care.
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Estimation of fetal weight by ultrasound

SUMMARY:
The purpose of this randomized controlled trial is to compare the frequency of the diagnosis of fetal growth abnormalities when ultrasound assessment is performed at 2 versus 4 week intervals.

DETAILED DESCRIPTION:
While there is an agreement that women at risk for abnormalities of fetal growth should have serial ultrasound examinations in the 3rd trimester, there is a lack of consensus on how frequently these exams should be done. The American College of Obstetrics and Gynecology recommend that an ultrasound to assess fetal growth be performed between 2 to 4 weeks; however, there have been no prospective or randomized trials to determine whether the optimal interval should be closer to 2 weeks or delayed to 4 weeks. Currently, only 60% of fetuses' with abnormal growth are detected antenatally. There is equipoise of whether ultrasound every 2 versus 4 weeks improves the detection and subsequent newborn outcomes or merely leads to an increase in false positives and unnecessary interventions. It has been proposed, that if delivery occurs within 2 weeks of the ultrasound, the antenatal detection of abnormal growth may be more accurate and hence more likely to improve outcomes. Conversely, a shorter interval may result in confusion as to whether there is actual change in growth or merely variation in the measurement technique itself. Moreover, with the cost of ultrasound averaging approximately $200 per examination, the interval between ultrasounds can have major implications on public-health costs as well as the interventions that subsequently follow if an abnormality is detected.

The purpose of this randomized controlled trial is to compare the frequency of the diagnosis of fetal growth abnormalities when ultrasound assessment is performed at 2 versus 4 week intervals.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age ≥ 18 years
* Singletons
* Gestational age ≥ 20 weeks to 27 weeks 6 days
* Has insurance, whether private or government issued
* High-risk pregnancy requiring serial fetal growth assessment as determined by the treating physician.
* Dating of pregnancy by ultrasound ≤ 21 weeks and 6 days of gestation or known date of conception in the setting of in vitro fertilization
* No known major anomalies

Exclusion Criteria:

* Known major fetal anomaly
* Multiple gestation (twins or triplets)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 228 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Frequency of detection of fetal growth abnormalities, starting at 28 weeks gestational age | up to 72 hours after delivery

SECONDARY OUTCOMES:
Birthweight compared to antenatal estimated fetal weights | At delivery
  Comparison of estimated fetal weight by ultrasound to actual birth weight at delivery
Frequency of detection of amniotic fluid abnormality, starting at 28 weeks gestational age | Up to 72 hours after delivery
Cost of interventions resulting from detection of abnormal growth or amniotic fluid | up to 72 hours from neonatal discharge from hospital
  e.g. additional ultrasounds, antenatal testing, hospital admission, induction, antepartum or intrapartum complications
Composite neonatal morbidity (CNM) | up to 72 hours from neonatal discharge from hospital
Composite maternal morbidity (CMM) | up to 72 hours from mother's discharge from hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Memorial Hermann Hospital, Texas Medical Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No